CLINICAL TRIAL: NCT03980821
Title: A Phase I, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AZD4635 in Japanese Patients With Advanced Solid Malignancies.
Brief Title: A Phase I Study of AZD4635 in Japanese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D8730C00005
Record Dates: First submitted 2019-05-24; First posted 2019-06-10 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Advanced Solid Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD4635 monotherapy (Experimental): Dose escalation of AZD4635 monotherapy for patients with advanced solid malignancies
  Interventions: Drug: AZD4635

INTERVENTIONS:
Drug: AZD4635 — AZD4635 taken orally

SUMMARY:
This is a Phase I, open-label study to assess the safety, tolerability, pharmacokinetics and anti-tumor activity of AZD4635 in Japanese patients with advanced solid malignancies. This study consists of 2 cohorts, Cohort1 and Cohort2. At least 3 or up to 6 evaluable Japanese patients with advanced solid malignancies will be enrolled in Cohort1 and 6 evaluable patients will be enrolled in Cohort2.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

Investigate the safety and tolerability of AZD4635 monotherapy in Japanese patients

Secondary objective:

Characterize the single-dose and multiple-dose plasma pharmacokinetic (PK) parameters of AZD4635 monotherapy Determine the preliminary anti-tumor activity of AZD4645 monotherapy

Overall design:

This is a phase I, open-label study of AZD4635 in Japanese patients with advanced solid malignancies.

The study consists of 2 cohorts, Cohort 1 and Cohort 2. At least 3 or up to 6 evaluable Japanese subjects with advanced solid malignancies will be enrolled in Cohort 1 and 6 evaluable patients will be required for Cohort 2 to confirm the tolerability. The total number of evaluable subjects in each cohort will depend upon available data in each cohort and decision of Safety Review Committee(SRC).

Study Period:

The study is expected to start in June 2019 and end in June 2020.

Number of Subjects:

9 to 12 evaluable subjects will be enrolled in this study to confirm the tolerability.

Treatments and treatment duration:

Subjects will receive AZD4635 once daily (QD). A single dose of AZD4635 will be taken on Cycle 0 Day1 and the subsequent dose of AZD4635 will be taken from Cycle 1 Day 1 until discontinuation criterion is met. A cycle of study treatment will be defined as 21 days of continuous dosing.

ELIGIBILITY:
Major Inclusion Criteria:

* Adult subjects; age ≥ 20 years
* Histologically or cytological confirmation of a solid, malignant tumor, excluding central nervous system (CNS) tumors and lymphoma, that is refractory to standard therapy or for which no standard of care regimen currently exists
* Patients must have either at least one lesion that can be evaluable using RECIST v1.1 or patients with mCRPC must have measurable prostate specific antigen above normal limits (per local ranges)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Normotensive or well controlled blood pressure, with or without current antihypertensive treatment
* Females of child-bearing potential must use 2 highly effective methods of contraception
* Male patients should be willing to use barrier contraception

Major Exclusion Criteria:

* Any investigational medicinal product or other systemic anticancer treatment within at least 4 weeks prior to the first dose of study treatment, or within 8 weeks after immunotherapy or other long half-life antibody therapy, whichever is the most appropriate and as judged by the Investigator.
* Evidence of recent or significant cardiovascular disease
* Unresolved toxicities from prior therapy greater than CTCAE Grade 1 at starting study treatment
* History of seizures, CNS tumors or CNS metastasis
* Active or prior documented autoimmune or inflammatory disorders within the past 3 years to the start of treatment
* Patients with prior ≥ Grade3 immune-mediated reactions
* Evidence of severe or uncontrolled systemic diseases
* Inadequate bone marrow reserve or organ function
* Refractory nausea and vomiting, chronic gastrointestinal diseases, or previous significant bowel resection that would preclude adequate absorption of AZD4635
* History of hypersensitivity to AZD4635 or drugs with a similar chemical structure or class to AZD4635
* Judgment by the Investigator that the patient should not participate in the study

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
The incidence of Adverse event and SAE | From the informed consent to 30 days post last dose
  Investigate the safety and tolerability of AZD4635
The incidence of Dose-limiting toxicity (DLTs) | 25 days (Cycle0 and Cycle1)
  Investigate the safety and tolerability of AZD4635

SECONDARY OUTCOMES:
Objective response rate (ORR) | Tumor assessment is Cycle 4 Day 1 and then on Day 1 of each even numbered cycle (+/-5 days) until disease progression. Expected to be for up to 6 months.
  Summarize based on RECIST 1.1 by cohort and overall.
Maximum plasma concentration (Cmax) | Samples will be collected at pre-specified time points in the single-dose and multiple-dose portion of the study beginning with Cycle 1 Day 1 until last dose. Expected to be for up to 6 months.
  Characterize the single-dose and multiple-dose plasma of AZD4635
Disease control rate (DCR) | Tumor assessment is Cycle 4 Day 1 and then on Day 1 of each even numbered cycle (+/-5 days) until disease progression. Expected to be for up to 6 months.
  Summarize based on RECIST 1.1 by cohort and overall.
Area under the plasma concentration-time curve (AUC) | Samples will be collected at pre-specified time points in the single-dose and multiple-dose portion of the study beginning with Cycle 1 Day 1 until last dose. Expected to be for up to 6 months.
  Characterize the single-dose and multiple-dose plasma of AZD4635

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Matsubara N, Kusuhara S, Yamamoto N, Sudo K, Yanagita M, Murayama K, Kawasumi H, Russell DL, Yin D, Shimizu T. Safety and pharmacokinetics of imaradenant (AZD4635) in Japanese patients with advanced solid malignancies: a phase I, open-label study. Cancer Chemother Pharmacol. 2024 Apr;93(4):341-352. doi: 10.1007/s00280-023-04605-9. Epub 2023 Dec 13. PMID 38086998